CLINICAL TRIAL: NCT07145203
Title: Effect of Virtual Reality on Anxiety, Stress, Pain and Patient's Satisfaction Among Palestinian Patients Undergoing Colonoscopy: A Randomized Controlled Trial
Brief Title: Virtual Reality on Anxiety, Stress, Pain and Patient's Satisfaction Among Patients Undergoing Colonoscopy
Acronym: VR/RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, khulud "Mohammad Hasham" Hasham Mansor, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB R-2024/A/129/N
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Stress; Pain; Patient Satisfaction; Patients Undergoing Colonoscopy
Keywords: Virtual Reality; Anxiety; Stress; Pain; Patient Satisfaction; Palestinian Patients; Colonoscopy
MeSH Terms: conditions — Anxiety Disorders; Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Participants in the VR group wore a VR headset during the colonoscopy procedure, while the control group received standard care without VR.
  The intervention used the Guided Meditation VR application developed by Cubicle Ninjas Agency, featuring immersive 360-degree natural environments such as tropical beach, diving, forests, and snowy landscapes. Patients chose one environment accompanied by relaxing music and nature sounds.
  VR sessions lasted 15 to 30 minutes during the colonoscopy, with the headset worn to immerse patients in the selected environment. The session was stopped if the patient experienced discomfort or requested removal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): The VR intervention utilized a head-mounted VR headset with built-in headphones. Patients selected VR environments from a predefined list of natural scenes, including tropical beach, diving, forest, and snowy landscape, each accompanied by relaxing music and nature sounds. The Guided Meditation VR application from Cubicle Ninjas (https://guidedmeditationvr.com/) provided 360-degree immersive nature environments with standardized calming background audio. VR was applied during the colonoscopy procedure, with sessions lasting 15 to 30 minutes and discontinued if the patient experienced nausea, dizziness, or requested removal.
  Interventions: Device: Meta Quest 2 VR headset
- control group (No Intervention): Participants in the control group received only standard care according to the hospital's protocol during the colonoscopy procedure.

INTERVENTIONS:
Device: Meta Quest 2 VR headset — The VR intervention used a head-mounted VR headset with built-in headphones. Patients selected VR environments from a predefined list of four nature scenes (tropical beach, diving, forest, and snowy landscape) with relaxing music and nature sounds. Guided Meditation VR from Cubicle Ninjas (https://guidedmeditationvr.com/) featured 360-degree immersive nature environments with standardized calming background audio. VR was applied during the colonoscopy procedure, with sessions lasting 15 to 30 minutes and discontinued if the patient reported nausea, dizziness, or requested removal.
  Arms: VR group

SUMMARY:
The goal of this randomized controlled trial was to investigate the effect of Virtual Reality (VR) on anxiety, stress, pain, and patient satisfaction among Palestinian patients undergoing colonoscopy. The study aimed to determine the efficacy of VR as a non-pharmacological intervention to improve the patient experience during the procedure.

The main research hypotheses are:

H01: There will be no significant difference in anxiety levels between patients who receive immersive VR during colonoscopy and those who receive standard care.

H02: There will be no significant difference in perceived stress levels between patients who receive immersive VR during colonoscopy and those who receive standard care.

H03: There will be no significant difference in pain levels between patients who receive immersive VR during colonoscopy and those who receive standard care.

H04: There will be no significant difference in satisfaction levels between patients who receive immersive VR during colonoscopy and those who receive standard care.

Participants will:

Receive either a VR intervention or standard care during their colonoscopy. Wear a VR headset for 15-30 minutes, immersing themselves in a natural environment with relaxing music and nature sounds.

Complete assessments of anxiety, stress, pain, and satisfaction before and after the procedure using validated questionnaires.

DETAILED DESCRIPTION:
Title: Effect of Virtual Reality on Anxiety, Stress, Pain, and Patient Satisfaction among Palestinian Patients Undergoing Colonoscopy: A Randomized Controlled Trial

Background: Colonoscopy is a common diagnostic and therapeutic procedure for gastrointestinal disorders but often causes anxiety, stress, and pain, which can complicate the procedure and increase sedative use. Virtual reality (VR) technology offers immersive, multi-sensory environments that may reduce these negative psychological and physical responses. This study aims to evaluate the effect of VR on anxiety, stress, pain, and patient satisfaction among Palestinian patients undergoing colonoscopy.

Methods: A randomized controlled trial will be conducted at the Endoscopy Unit of Rafidia Surgical Hospital in Nablus, Palestine. A total of 150 patients scheduled for colonoscopy will be randomly assigned to either the VR group (n=75) or the control group (n=75). The VR group will wear head-mounted VR devices for 15 to 30 minutes during the procedure, choosing from natural environments such as tropical beaches, forests, or snowy landscapes accompanied by relaxing music and nature sounds. Data on anxiety, stress, pain, and satisfaction will be collected through questionnaires administered by the researcher. The study duration is three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective colonoscopy
* Patients older than 18 years
* Patients with no history of previous colonoscopy procedures
* Patients experiencing moderate to severe anxiety and stress

Exclusion Criteria:

* Patients who have a history of psychiatric disorders, epilepsy, hypertension, or chronic pain.
* Patients who are mute and could not read, or write, patients with visual, hearing, or cognitive impairment.
* Patients who implanted hearing aids or cardiac pacemakers.
* Patients who were given any anxiolytic, sedative, or hypnotic drugs before or during procedure.
* Patients who were exposed to complications during the operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | before colonoscopy and then 60 minutes post-procedure
  The STAI score ranges between 20-80, the higher score indicating greater anxiety. It is classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80)
Perceived Stress Scale (PSS-10) | before colonoscopy and then 60 minutes post-procedure
  The PSS-10 score can range from 0 to 40 with higher scores indicating higher perceived stress. It is classified as "no or low anxiety" (0-13), "moderate anxiety" (14-26), and "high anxiety" (27-40).

CONTACTS AND LOCATIONS:
Locations (1):
- Rafidia Surgical Governmental Hospital, Nablus, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) cannot be shared due to ethical concerns about participant privacy and the inappropriate use of data. Also, compliance with journal publication policies.

REFERENCES:
- See also: the website Guided Meditation VR application, developed by Cubicle Ninjas Agency — https://guidedmeditationvr.com/